CLINICAL TRIAL: NCT07039552
Title: Development and Validation of an Ovarian Cancer Risk Prediction Model for Family Members of Ovarian Cancer Probands With BRCA1/2 Germline Mutations
Brief Title: Development and Validation of an Ovarian Cancer Risk Prediction Model for Family Members of Ovarian Cancer Probands
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Tengyun HOC
Record Dates: First submitted 2025-05-28; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-04

CONDITIONS: Hereditary Breast and Ovarian Cancer Syndrome; BRCA Mutations
Keywords: BRCA1 or BRCA2 germline mutations; hereditary ovarian cancer
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Participants in this study will have 4ml of peripheral blood collected for genetic testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Members of ovarian cancer families carrying BRCA1/2 germline mutations: Members of ovarian cancer families carrying BRCA1/2 germline mutations，telephone follow-ups will be conducted once a year to longitudinally monitor ovarian cancer incidence and to collect diagnostic evidence.
  Interventions: Procedure: risk-reducing salpingo-oophorectomy (RRSO)

INTERVENTIONS:
Procedure: risk-reducing salpingo-oophorectomy (RRSO) — The proportion of BRCA1/2 germline mutation carriers in the high-risk population of ovarian cancer who undergo risk-reducing salpingo-oophorectomy (RRSO). RRSO refers to the preventive surgical removal of both fallopian tubes and ovaries to reduce the risk of ovarian cancer, fallopian tube cancer, and peritoneal cancer.

SUMMARY:
Ovarian cancer is the gynecological malignancy with the highest fatality rate, seriously threatening the life and health of women. One of the main reasons for its high fatality rate is that approximately 70% of patients are diagnosed at an advanced stage. Fortunately, about 1/5 of ovarian cancers are associated with genetic factors, providing us with an opportunity to screen high-risk populations and thereby prevent and diagnose the disease at an early stage and reduce the disease burden.

Currently, research related to hereditary ovarian cancer in China is still very scarce, and clinical practice relies on data from foreign studies. However, hereditary tumors have distinct regional and ethnic characteristics, making it urgent to conduct clinical research based on the Chinese population to guide clinical practice in China. Current research suggests that approximately 50% - 60% of hereditary ovarian cancers are closely related to the BRCA1/2 genes. Therefore, accurately assessing the risk of ovarian cancer in BRCA1/2 germline mutation carriers is of great significance for the prevention and treatment of hereditary ovarian cancer.

DETAILED DESCRIPTION:
This study will adopt a multicenter ambispective cohort study design to comprehensively collect and analyze the clinical characteristics, family characteristics, gene mutation characteristics, and lifestyle data of BRCA1/2 germline mutation carriers. For family members who have not yet developed ovarian cancer at the time of enrollment, telephone follow-ups will be conducted once a year to longitudinally monitor ovarian cancer incidence and to collect diagnostic evidence.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed with ovarian malignant tumor.

  * Identified as carriers of BRCA1/2 germline pathogenic or likely pathogenic mutations through genetic testing, in accordance with the "Standards and Guidelines for the Interpretation of Sequence Variants" (2015 Edition) of the American College of Medical Genetics and Genomics (ACMG).

    * Age of 18 years or older. ④ Voluntary participation in this research and signing of the informed consent form.

Exclusion Criteria:

* ① Patients who refuse to provide necessary information.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women can develop ovarian cancer
Study Population: This study will adopt a multicenter ambispective cohort study design to comprehensively collect and analyze the clinical characteristics, family characteristics, gene mutation characteristics, and lifestyle data of BRCA1/2 germline mutation carriers. For family members who have not yet developed ovarian cancer at the time of enrollment, telephone follow-ups will be conducted once a year to longitudinally monitor ovarian cancer incidence and to collect diagnostic evidence.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2035-12-30 (Estimated)

PRIMARY OUTCOMES:
The age at which pathologically diagnosed with ovarian malignant tumors (ICD-10 C56) | From enrollment to the end of follow-up at 5 years
  The age at which pathologically diagnosed with ovarian malignant tumors (ICD-10 C56)

SECONDARY OUTCOMES:
Acceptance rate of risk-reducing salpingo-oophorectomy (RRSO) among BRCA1/2 mutation carriers | From enrollment to the end of follow-up at 5 years
  The proportion of BRCA1/2 germline mutation carriers in the high-risk population of ovarian cancer who undergo risk-reducing salpingo-oophorectomy (RRSO). RRSO refers to the preventive surgical removal of both fallopian tubes and ovaries to reduce the risk of ovarian cancer, fallopian tube cancer, and peritoneal cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-19): https://cdn.clinicaltrials.gov/large-docs/52/NCT07039552/Prot_SAP_ICF_000.pdf